CLINICAL TRIAL: NCT06143774
Title: A Phase I, Open-label, Dose-finding Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of TRX-920 Oral Gel (10 mg and 30 mg) in Patients With Advanced Solid Tumors
Brief Title: Study of TRX-920 for Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TaiRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNOF-001
Record Dates: First submitted 2023-11-06; First posted 2023-11-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor
Keywords: TRX-920 Oral Gel; SN38

STUDY DESIGN:
Intervention Model Description: Dose-finding Study using 3+3 design.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TRX-920 Oral Gel (Experimental): Dose escalation (escalation from 1, 2, 4, 8, 16, 30, 60, 90 mg TRX-920 Oral Gel)
  Interventions: Drug: TRX-920 Oral Gel (10 mg and 30 mg)

INTERVENTIONS:
Drug: TRX-920 Oral Gel (10 mg and 30 mg) — TRX-920 Oral Gel will be administered orally at a week (BIW) in an 8-week cycle. No food should be taken 2 hours before and 1 hour after taking TRX-920. The dose escalation/de-escalation rules will be based on definitions of dose-limiting toxicity (DLT) and will be monitored during the first treatment cycle (i.e., the first 4 weeks post the first dose).
  The starting dose will be 1 mg and the dosing frequency is twice every week (BIW). Subjects will be assigned to a dose level in sequential cohorts based on the order of their enrollment. The dose escalation will follow a 3+3 design and doses escalate from approximately 1 mg BIW, 2 mg BIW, 4 mg BIW, 8 mg BIW, and 16mg BIW and the doses for subsequent cohorts will be determined by Safety Review Committee (SRC). Dose escalation will be stopped till the maximum tolerated dose (MTD) is reached or identified.

SUMMARY:
The study drug TRX-920 Oral Gel contains SN38, an active metabolite of Irinotecan (CPT-11), which is a widely prescribed anti-cancer drug that has been approved in many countries for the treatment of colorectal and pancreatic cancer. TRX-920 is the oral gel formulation that directly contains SN38 instead of Irinotecan. A series of biology and animal studies have demonstrated that the TRX-920 Oral Gel could inhibit tumor growth with fewer side effects compared to Irinotecan.

DETAILED DESCRIPTION:
This is the first study in which the study drug TRX-920 Oral Gel is being given to humans. However, as a metabolite of Irinotecan, SN38 has proved its effectiveness in the treatment of colorectal and pancreatic cancer. TRX-920 also showed its effect of anti-tumor in various cancer cell lines and animal models. The purposes of this study are to find the highest dose of the study drug that can be given without causing significant side effects, the side effect of the study drug, the concentration of the study drug in the blood, and the effect on your specific cancer.

The clinical study will be conducted in Taiwan. The drug used in this study is an investigational product (TRX-920 Oral Gel) which is provided free of charge by TaiRx, Inc. (a pharmaceutical company in Taiwan, and is the sponsor of this study), and is a potential oral anti-cancer therapy for patients suffering from various cancers.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for enrollment in the study:

1. Signed and dated informed consent form
2. Histologically and cytologically confirmed advanced solid tumor malignancies that are refractory to standard therapy or have no accepted standard therapy.
3. Solid tumors that are measurable or evaluable as per Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Target lesions that have been previously irradiated will not be considered measurable (lesion).
4. Female or male, 18 years of age or older.
5. ECOG performance status 0 or 1.
6. QTcF ≤ 480 ms at screening.

Exclusion Criteria:

1. Patients with homozygous or compound heterozygous genotypes for UGT1A1*28 and *6 alleles (e.g., *28/*28, *6/*6, *6/*28).
2. Clinically significant comorbidity such as unstable angina, congestive heart failure (NYHA Grade III or IV), uncontrolled hypertension (>160/100 mmHg despite optimal medical treatment), chronic obstructive pulmonary disease (COPD) with frequent exacerbations, refractory asthma, inflammatory bowel disease or intestinal obstruction.
3. Acute myocardial infraction or cerebrovascular accident (CVA) within 6 months prior the first dose of study drug.
4. Central nervous system (CNS) metastasis or seizure disorder due to underlying malignancy except those who have been treated and have stable CNS metastases or are asymptomatic.
5. AIDS-defining opportunistic infections within the past 12 months.
6. HBV infection (positive HBsAg) except for carrier of inactive HBV as defined by negative HBeAg with normal ALT and HBV DNA < 2,000 IU/mL or HCV infection (positive anti-HCV antibody) except for those with undetectable HCV RNA.
7. Inadequate bone marrow reserve, hepatic or renal function as defined by any of the following laboratory values:

   1. absolute neutrophil count (ANC) < 1500/µL
   2. platelet count < 90,000/µL
   3. hemoglobin < 9 g/dL
   4. total bilirubin > 1.5*the upper limit of normal (ULN)
   5. aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3*ULN if no hepatic metastases are present; > 5*ULN if hepatic metastases are present
   6. Non-indexed eGFR < 60 mL/min (formula in Appendix 4)
8. Toxicities resulting from prior therapy or surgical procedures not yet resolved to ≤ NCI CTCAE v5.0 Grade 1 with the exception of alopecia, skin hyperpigmentation or hypopigmentation or grade 2 toxicity with prior approval of the Medical Monitor.
9. Major surgical procedures (as defined by Investigator) within 4 weeks prior to the first dose of study drug or any ongoing post-operative complications.
10. Receiving any radiotherapy within 3 months
11. Receiving any (investigational or approved) anti-cancer therapy (including chemotherapy or targeted therapy) within 28 days or 5 half-lives (whichever is longer) prior to the first dose of study drug
12. A history of apparent allergic reactions to irinotecan injection (dosed with prior treatment with prophylactic drug)
13. If female, is pregnant or breastfeeding
14. If men or women with childbearing potential, unwilling to use effective contraceptive methods during the study and for at least 3 months (men) or 1 month (women) after the last dose of study drug. Effective contraceptive methods include implants, injectables, combined oral contraceptives, intra-uterine devices (IUDs), sexual abstinence, surgical sterilization, or a partner who is sterile.
15. Receiving live attenuated vaccine within 28 days prior to the first dose of study drug.
16. Life expectancy < 3 months.
17. Other prior or ongoing condition(s) that, in the opinion of the investigator, could affect the safety of the subject, compromise the subject's ability to comply with the study requirements or impair the assessment of study results.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) of TRX-920 Oral Gel | the first 4 weeks post the first dose
  The MTD is defined as the highest dose level at which no more than 1 in 6 subjects experiences a DLT. The recommended Phase 2 dose (RP2D) will be determined by Safety Review Committee based on all available PK, safety, and preliminary efficacy data. The RP2D will not exceed the MTD.
Frequency, type, severity and relationship to study drug of adverse events (AEs) of TRX-920 Oral Gel | Cycle 1 Day 1 to study completion, an average of 1 year (each cycle is 56 days)
  AEs will be coded by system organ class (SOC) and preferred term according to the Medical Dictionary for Regulatory Activities (MedDRA) system.

SECONDARY OUTCOMES:
Drug exposure and human pharmacokinetics (Cmax) of SN38 derived from plasma concentration-time profiles | Cycle 1 Day 1 to study completion, an average of 1 year (each cycle is 56 days)
  The plasma concentrations of SN38 will be analyzed using compartmental or non-compartmental approach to calculate Cmax for individual subjects.
Drug exposure and human pharmacokinetics (Tmax) of SN38 derived from plasma concentration-time profiles | Cycle 1 Day 1 to study completion, an average of 1 year (each cycle is 56 days)
  The plasma concentrations of SN38 will be analyzed using compartmental or non-compartmental approach to calculate Tmax for individual subjects.
Drug exposure and human pharmacokinetics (MRT) of SN38 derived from plasma concentration-time profiles | Cycle 1 Day 1 to study completion, an average of 1 year (each cycle is 56 days)
  The plasma concentrations of SN38 will be analyzed using compartmental or non-compartmental approach to calculate MRT for individual subjects.
Drug exposure and human pharmacokinetics (AUC) of SN38 derived from plasma concentration-time profiles | Cycle 1 Day 1 to study completion, an average of 1 year (each cycle is 56 days)
  The plasma concentrations of SN38 will be analyzed using compartmental or non-compartmental approach to calculate AUC for individual subjects.
Drug exposure and human pharmacokinetics (terminal half-life) of SN38 derived from plasma concentration-time profiles | Cycle 1 Day 1 to study completion, an average of 1 year (each cycle is 56 days)
  The plasma concentrations of SN38 will be analyzed using compartmental or non-compartmental approach to calculate terminal half-life (T 1/2) for individual subjects.
Objective response rate (ORR) per RECIST v1.1 | Cycle 1 Day 1 to study completion, an average of 1 year (each cycle is 56 days)
  Tumor assessment by computed tomography (CT) or magnetic resonance imaging (MRI) will be performed every 8-week cycle starting from Cycle 2 Day 1. All subjects will attend an End of Treatment (EOT) visit at the time decision is made to discontinue study drug administration.
  The Objective response rate (ORR) as per RECIST v1.1 will be calculated in the efficacy population.
Disease control rate (DCR) per RECIST v1.1 | Cycle 1 Day 1 to study completion, an average of 1 year (each cycle is 56 days)
  Tumor assessment by computed tomography (CT) or magnetic resonance imaging (MRI) will be performed every 8-week cycle starting from Cycle 2 Day 1. All subjects will attend an End of Treatment (EOT) visit at the time decision is made to discontinue study drug administration.
  The disease control rate (DCR) as per RECIST v1.1 will be calculated in the efficacy population.
Duration of response (DOR) per RECIST v1.1 | Cycle 1 Day 1 to study completion, an average of 1 year (each cycle is 56 days), assessed up to 24 months
  Tumor assessment by computed tomography (CT) or magnetic resonance imaging (MRI) will be performed every 8-week cycle starting from Cycle 2 Day 1. All subjects will attend an End of Treatment (EOT) visit at the time decision is made to discontinue study drug administration.
  The duration or response (DOR) as per RECIST v1.1 will be calculated in the efficacy population.
Time to tumor progression (TTP) per RECIST v1.1 | Cycle 1 Day 1 to study completion, an average of 1 year (each cycle is 56 days), assessed up to 24 months
  Tumor assessment by computed tomography (CT) or magnetic resonance imaging (MRI) will be performed every 8-week cycle starting from Cycle 2 Day 1. All subjects will attend an End of Treatment (EOT) visit at the time decision is made to discontinue study drug administration.
  The time to tumor progression (TTP) as per RECIST v1.1 will be calculated in the efficacy population.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Yuan Bai, M.D., Principal Investigator — China Medical University, Taiwan
Locations (3):
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - Taipei Medical University Hospital, Taipei